CLINICAL TRIAL: NCT05888025
Title: A Pilot Proof of Concept, Single-Center Study of the Effects of Telephone-Delivered Mindfulness-based Cognitive Therapy (MBCT-T) on Preoperative Pain Catastrophizing and Pain Outcomes After Spine Surgery
Brief Title: MBCT-T for Preoperative Pain Catastrophizing and Pain Outcomes After Spine Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporarily suspended.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00339
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBCT-T (Experimental): Participants with high pain catastrophizing who are scheduled for spine surgery will receive four weekly sessions of preoperative telephone-delivered mindfulness-based cognitive therapy (MBCT-T). They will then be followed for two weeks postoperatively.
  Interventions: Behavioral: Telephone-Delivered Mindfulness-based Cognitive Therapy (MBCT-T)

INTERVENTIONS:
Behavioral: Telephone-Delivered Mindfulness-based Cognitive Therapy (MBCT-T) — MBCT-T will be delivered in groups of four to eight subjects by telephone using a conference line with NYULH WebEx. Participants will receive a workbook containing session content and home practice logs and audio guides for home practice. Subjects will complete individual orientation sessions with the MBCT-T facilitator prior to start of the group sessions. The four subsequent weekly group sessions are approximately 90 minutes long. Participants will be encouraged to practice daily meditation in between group sessions for 20-30 minutes, six days per week

SUMMARY:
This is a two phase study. In phase 1, a focus group (N=5) will be conducted to adapt MBCT-T for use in the study population. In phase 2, a single-arm trial will be conducted examining four, weekly sessions of preoperative MBCT-T in subjects with high pain catastrophizing scheduled for spine surgery (N=20). Subjects will then be followed for two weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for one or two level lumbar spine surgery requiring an inpatient stay as well as patients having ambulatory 1 or 2 level lumbar spine surgeries
* PCS score ≥ 20
* Able to provide voluntary informed consent
* Telephone access
* Internet access

Exclusion Criteria:

* Non-English speaking
* Cognitively impaired, by history
* Bipolar disorder
* Borderline personality disorder
* Active post-traumatic stress disorder
* Schizoaffective disorder or any other disorder characterized by delusions or hallucinations
* History of self-harm or suicidality in past three months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Attend More than Half of Scheduled Sessions | Up to Week 8 (End of Intervention)
Client Satisfaction Questionnaire (CSQ-8) Score | Week 8 (End of Intervention)
  The CSQ-8 is an 8-item questionnaire assessing satisfaction with the intervention. Each item is rated on a 4-point scale from 1-4. The total score is the sum of responses and ranges from 8 to 32, with the higher number indicating greater satisfaction.

SECONDARY OUTCOMES:
Change in Pain Catastrophizing Scale (PCS) Score | Baseline, Week 8
  The PCS is a 13-item questionnaire designed to quantify an individual's pain experience, asking about how they feel and what they think about when they are in pain. Each item is rated on a 5-point scale ranging from 0 (not at all) to 4 (all the time). The total score is the sum of responses and ranges from 0 to 52. Higher scores represent greater pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Doan, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, Brooklyn, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: lisa.doan@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to lisa.doan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.